CLINICAL TRIAL: NCT00605904
Title: Modulation of Pharmacologically Induced Alcohol Craving in Recently Detoxified Alcoholics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Markus Heilig, Clinical Director, NIAAA, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 080058; 08-AA-0058 (Other: NIH)
Record Dates: First submitted 2008-01-30; First posted 2008-01-31 (Estimated); Results first posted 2012-07-03 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-05

CONDITIONS: Alcoholism
Keywords: Chemical Stressor; Alcoholism; Yohimbine; Acamprosate; Craving
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate; Yohimbine; 6-chloro-2-(1-piperazinyl)pyrazine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acamprosate (Experimental): Subjects received 3 tablets of 333mg acamprosate orally, three times daily (total dose of 999 mg) for a minimum of 2 weeks.
  Interventions: Drug: Acamprosate; Drug: Yohimbine; Drug: mCPP; Drug: Saline
- Placebo (Placebo Comparator): Subjects received 3 tablets of placebo orally, three times daily, for a minimum of 2 weeks.
  Interventions: Drug: Yohimbine; Drug: mCPP; Drug: Saline

INTERVENTIONS:
Drug: Acamprosate — orally administered tablet, 333mg, three times daily for a minimum of 2 weeks (14 days)
  Other Names: Campral
  Arms: Acamprosate
Drug: Yohimbine — Intravenous infusion of yohimbine (0.4 mg/kg) administered once over 10 minutes
  Other Names: Yohimbe; Yocon; Yohimex; Aphrodyne
Drug: mCPP — Intravenous infusion of mCPP (0.05 mg/kg) over 10 minutes, two times, for a total of 0.1 mg/kg
  Other Names: 3-CPP; CPP
Drug: Saline — Intravenous infusion of 0.9% sodium chloride solution over 10 minutes, three times during the study (2 times for the "Saline Infusion" milestone, and one time immediately following the "Yohimbine Infusion" milestone)
  Other Names: Normal Saline Flush; Sodium Chloride

SUMMARY:
This study will determine if acamprosate, a drug approved to treat alcoholism, decreases alcohol cravings in alcohol-dependent subjects following infusions of yohimbine and mCPP. Yohimbine causes anxiety and may provoke a desire for alcohol; mCPP induces a feeling of having had a few drinks, which often creates a desire for more drinks. If acamprosate can prevent a craving following these stimuli, then the effectiveness of new experimental drugs for treating alcoholism can be tested for their ability to block yohimbine or mCPP-induced cravings. This type of investigation would be less expensive and less time-consuming than conducting clinical trials with alcohol-dependent people.

People between 21 and 65 years of age who are alcohol-dependent and have been drinking regularly for at least 1 month before entering the study may be eligible to participate.

Participants are admitted to the NIH Clinical Center for about 35 days, during which time they are asked to participate in an alcohol treatment program. They may request passes to leave the hospital during the day but must return overnight. Upon return to the hospital, subjects are required to take a breathalyzer test for alcohol and urine screen for drug use. Participants found to have used drugs or consumed alcohol while away from the hospital are terminated from the study.

Participants are randomly assigned to take acamprosate or placebo pills three times a day for about 2 weeks. They are then given three intravenous (through a vein) infusions, 5 to 7 days apart, each containing either yohimbine, mCPP or placebo. The drugs are infused for 20 minutes following a 1-hour infusion of saline (salt water). Subjects complete two questionnaires - an alcohol urge questionnaire to assess the desire for alcohol and a PASS rating scale to assess anxiety - several times during the study and during the infusions....

DETAILED DESCRIPTION:
Objective: The objective of the present study is to establish, in our laboratory, a published model of pharmacologically induced alcohol craving, and carry out an initial evaluation of its predictive validity for efficacy in treatment of alcoholism. Two pharmacological challenges are tested: 1. The alpha2-adrenergic antagonist yohimbine, which reliably induces reinstatement of alcohol seeking in experimental animals, but has produced less clear results in humans. 2. The serotonergic compound mCPP, which has been reported to robustly increase alcohol craving in human alcoholics, but for which animal data are less clear. Our objective study is to evaluate craving responses to infusion of yohimbine or mCPP using optimal assessment tools and subject population, and establish their sensitivity to the clinically effective alcoholism medication acamprosate.

Study Population: The study will be carried out in 60 subjects aged 21-65 years, with alcohol dependence as their primary complaint, and without other serious medical or psychiatric conditions. An additional inclusion criterion will be elevated trait anxiety as measured by the Spielberger Trait Anxiety Inventory. Subjects will be admitted to the NIAAA research inpatient unit at the NIH Clinical Research Center (CRC) through the platform training and natural history protocol (05-AA-0121 Assessment and Treatment of People with Alcohol Drinking Problems ), which provides basic assessments and standard withdrawal treatment if needed. Patients will enter into the present protocol once such treatment, if needed, is completed.

Design: Following inclusion, subjects will be randomized to acamprosate (n=25) or placebo (n=25), receiving either 3 tablets of 333mg acamprosate three times daily, or receiving identically looking placebo. Following a minimum of 2 weeks of treatment, subjects will undergo three challenge sessions, a minimum of 5 days apart, with yohimbine, m-CPP or placebo infusion, in counterbalanced order.

Outcome Measures: During the challenge sessions, subjective cravings for alcohol will be assessed using the Alcohol Urge Questionnaire. Neuroendocrine and cardiovascular measures will be collected for exploratory purposes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be 60 recently detoxified alcoholics according to the following criteria:

* DSM-IV diagnosis of alcohol dependence on SCID, alcohol problems as primary complaint among substance use disorder, and alcohol use within the last month.
* Spielberger trait anxiety (21) score greater than 39
* Age 21-65
* Females of childbearing potential must agree to use a reliable method of birth control during the study. Reliable methods of birth control include oral contraceptives or Norplant(Registered Trademark); barrier methods such as diaphragms with contraceptive jelly, cervical caps with contraceptive jelly, condoms with contraceptive foam, or intrauterine devices; a partner with a vasectomy; or abstinence from intercourse.

EXCLUSION CRITERIA:

* People who present with significant medical problems which in the assessment of the Lead Associate Investigator contraindicate administration of any of the study drugs. Examples are patients requiring intensive medical or diagnostic management, such as uncontrolled hypertension, serious GI bleeding, major organ or body system dysfunction such as decompensated liver disease, renal failure, myocardial ischemia, congestive heart failure or cerebrovascular disease, major endocrine problems such as uncontrolled diabetes, pancreatic or thyroid disease, or glaucoma.
* People who are infected with the Human Immunodeficiency Virus (HIV).
* People with the following specific neuro-psychiatric disorders: any psychotic disorder including schizophrenia; bipolar affective disorder; or panic disorder.
* People with any other condition that impairs judgment or cognitive function to an extent that precludes them from providing informed consent or complying with treatment (incompetent individuals); or that requires management with pharmacotherapy that would make the subject ineligible for participation.
* Contraindications for acamprosate (previously exhibited hypersensitivity to acamprosate calcium or any of its components; or severe renal impairment, manifested as creatinine clearance of 30 mL/min or less.
* Contraindications for yohimbine or mCPP, such as liver or renal disease; chronic inflammation of the sexual organs or prostate gland; history of gastric and duodenal ulcers; glaucoma; hypersensitivity to yohimbine or mCPP
* People who are unlikely or unable to complete the treatment program because they become, or are likely to be, incarcerated while on the protocol.
* People who are required to receive treatment by a court of law or who are involuntarily committed to treatment.
* Pregnancy or lactation (negative pregnancy test required)
* Regular use of psychotropic medication, physician prescribed or purchased over the counter (e.g. antidepressant, lithium, antipsychotic, anxiolytic, antiepileptic, nasal decongestants in tablet form) or blood pressure medication (e.g. beta-blockers, calcium antagonists, ACE-inhibitors or AT1 antagonists) within the last 4 weeks, with the exception of benzodiazepines administered within the NIAAA program as part of alcohol withdrawal treatment. Specifically, no subject will be taken off psychoactive medications for the purpose of enrollment in this protocol.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Heilig M, Egli M. Pharmacological treatment of alcohol dependence: target symptoms and target mechanisms. Pharmacol Ther. 2006 Sep;111(3):855-76. doi: 10.1016/j.pharmthera.2006.02.001. Epub 2006 Mar 20. PMID 16545872
- [Background] Heilig M, Koob GF. A key role for corticotropin-releasing factor in alcohol dependence. Trends Neurosci. 2007 Aug;30(8):399-406. doi: 10.1016/j.tins.2007.06.006. Epub 2007 Jul 16. PMID 17629579
- [Background] Bohn MJ, Krahn DD, Staehler BA. Development and initial validation of a measure of drinking urges in abstinent alcoholics. Alcohol Clin Exp Res. 1995 Jun;19(3):600-6. doi: 10.1111/j.1530-0277.1995.tb01554.x. PMID 7573780

RESULTS

PARTICIPANT FLOW:
Groups:
- Acamprosate: Subjects received 3 tablets of 333mg acamprosate three times daily
- Placebo: Subjects received 3 tablets of placebo three times daily
Period: Baseline Data Collection and Dosing
Arm/Group | Acamprosate | Placebo
Started | 13 (While 37 subjects were enrolled in the protocol, only 34 were randomized to a study arm) | 21 (While 37 subjects were enrolled in the protocol, only 34 were randomized to a study arm)
Completed | 13 | 16
Not Completed | 0 | 5
Period: Infusion Sessions
Arm/Group | Acamprosate | Placebo
Started | 13 | 16
Saline Infusion | 13 | 14
mCPP Infusion | 12 | 13
Yohimbine Infusion | 12 | 15 (Milestones (infusions) were not received in the same order for each subjects so are not consecutive.)
Completed | 12 (Subjects who completed all three types of infusion (given in a different order for each subject)) | 13 (Subjects who completed all three types of infusion (given in a different order for each subject))
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acamprosate | Placebo | Total
Number analyzed (Participants) | 13 | 21 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 21 | 34
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 12 | 18 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 20 | 33
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 11 | 14
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Craving Rating in Response to Saline Infusion
Description: Alcohol craving was measured using the Penn Alcohol Craving Scale (PACS). It is a 5-item self-administered instrument that measures frequency, intensity, and duration of thoughts about drinking, along with ability to resist drinking. There is a single outcome score than ranges from 0 to 30, with 30 being the maximum amount of alcohol craving.
Time Frame: 180 minutes after the start of the infusion
Population: The analyses included only those subjects who completed all three types of infusions (saline, meta-Chlorophenylpiperazine, and yohimbine)
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 12 | 13
Units on a scale | 1.704 (0.715) | 1.766 (0.627)

2. Primary Outcome: Alcohol Craving Rating in Response to Meta-Chlorophenylpiperazine
Description: as for outcome 1
Time Frame: 180 minutes after the start of the infusion
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 12 | 13
Units on a scale | 3.460 (1.352) | 5.416 (1.185)

3. Primary Outcome: Alcohol Craving Rating in Response to Yohimbine Infusion
Description: as for outcome 1
Time Frame: 180 minutes after the start of the infusion
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 12 | 13
Units on a scale | 3.613 (1.140) | 3.606 (1.000)

ADVERSE EVENTS:
Arm/Group | Acamprosate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 11/12 | 9/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acamprosate (N=12) | Placebo (N=13)
Abnormal Dreaming (General disorders) | 5 | 5
Abundance of Energy (General disorders) | 6 | 7
Aggressiveness (General disorders) | 0 | 1
Agitation (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 2 | 3
Coughing Spells (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Decreased Interest in Sex (Reproductive system and breast disorders) | 1 | 6
Diarrhea (Gastrointestinal disorders) | 3 | 2
Dry Mouth (General disorders) | 1 | 3
Euphoria (General disorders) | 1 | 2
Feeling Down (Psychiatric disorders) | 1 | 2
Headaches (General disorders) | 3 | 1
Heart Racing (Cardiac disorders) | 1 | 1
Impaired Concentration (General disorders) | 2 | 2
Irritability (Psychiatric disorders) | 2 | 1
Lack of Appetite (Metabolism and nutrition disorders) | 1 | 0
Lack of Energy (General disorders) | 3 | 5
Mood Swings (Psychiatric disorders) | 1 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Nervousness (General disorders) | 0 | 2
Painful Erections (Reproductive system and breast disorders) | 0 | 1
Paranoid (Psychiatric disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Restlessness (General disorders) | 3 | 2
Sensation of Prickling (Skin and subcutaneous tissue disorders) | 1 | 1
Shakiness (General disorders) | 1 | 2
Skin Flushing (Skin and subcutaneous tissue disorders) | 0 | 1
Sleepiness (General disorders) | 6 | 7
Sleeplessness (General disorders) | 6 | 6
Stomach Ache (Gastrointestinal disorders) | 2 | 2
Tightening of Airways (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes